CLINICAL TRIAL: NCT01193998
Title: Analysis of the Impact of Using a Validated Diagnostic Prediction Model of Acute Heart Failure in the Emergency Department
Brief Title: Impact of Validated Diagnostic Prediction Model of Acute Heart Failure in the Emergency Department
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Principal Investigator, Brian Steinhart, Physician, Unity Health Toronto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 09-310
Record Dates: First submitted 2010-09-01; First posted 2010-09-02 (Estimated); Last update posted 2014-06-16 (Estimated); Status verified 2014-06

CONDITIONS: Dyspnea; Acute Heart Failure; Shortness of Breath
MeSH Terms: conditions — Dyspnea | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Clinician exposed to Model result (Active Comparator)
  Interventions: Other: Treatment as per model probability
- Clinician blinded to Model result (Experimental)
  Interventions: Other: Treatment as per usual care

INTERVENTIONS:
Other: Treatment as per model probability — Patients randomized to the arm where the clinician is exposed to the model results should be treated as per the model probability (i.e. if the model probability suggests AHF the clinician should treat for AHF).
  Arms: Clinician exposed to Model result
Other: Treatment as per usual care — Patients randomized to the arm where the clinician is blinded to the model results will undergo diagnostic tests and receive treatment as per the clinician's judgment and usual care standards.
  Arms: Clinician blinded to Model result

SUMMARY:
The purpose of this study is to evaluate a validated diagnostic prediction model in the appropriate diagnosis of Acute Heart Failure (AHF) in patients presenting at the emergency department with undifferentiated dyspnea.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Presentation to the ED with undifferentiated shortness of breath

Exclusion Criteria:

* Dyspnea of obvious cause, e.g. chest trauma, obvious clinical exacerbation of known chronic obstructive disease
* Obvious pulmonary edema in a patient with a known diagnosis of HF and recently admitted to hospital for HF
* Clinician does not plan to treat for AHF at all, but rather to pursue other causes of dyspnea (i.e., probability of AHF ≤ 20%)
* Clinician plans to treat for AHF and not to pursue other causes of dyspnea (i.e., probability of AHF ≥ 80%)
* Acute coronary syndrome within one month
* Chronic renal failure (serum creatinine ≥ 250 mol/l)
* Anticipated life expectancy < 6 months due to non-cardiovascular causes
* Participation in another interventional outcome trial
* Inability to obtain informed consent, including inability of patient to understand English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2010-09; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Comparison of diagnostic model versus clinical judgment in appropriate diagnosis of Acute Heart Failure in dyspneic emergency department patients | 60 days after patient presentation to the emergency department

SECONDARY OUTCOMES:
Determine if use of the diagnostic prediction model leads to cost savings and better health outcomes | From randomization until 60 days after patient presentation to the emergency department

CONTACTS AND LOCATIONS:
Overall Officials: Brian Steinhart, MD, Principal Investigator — Unity Health Toronto; David Mazer, MD, Principal Investigator — Unity Health Toronto; Gordon Moe, MD, Principal Investigator — Unity Health Toronto
Locations (3):
- Wayne State University, Detroit, Michigan, United States
- St. Michael's Hospital, Toronto, Ontario, Canada
- Waikato Hospital Cardiology Clinical Trials Unit, Waikato, New Zealand

REFERENCES:
- [Background] Januzzi JL Jr, Camargo CA, Anwaruddin S, Baggish AL, Chen AA, Krauser DG, Tung R, Cameron R, Nagurney JT, Chae CU, Lloyd-Jones DM, Brown DF, Foran-Melanson S, Sluss PM, Lee-Lewandrowski E, Lewandrowski KB. The N-terminal Pro-BNP investigation of dyspnea in the emergency department (PRIDE) study. Am J Cardiol. 2005 Apr 15;95(8):948-54. doi: 10.1016/j.amjcard.2004.12.032. PMID 15820160
- [Background] McCullough PA, Nowak RM, McCord J, Hollander JE, Herrmann HC, Steg PG, Duc P, Westheim A, Omland T, Knudsen CW, Storrow AB, Abraham WT, Lamba S, Wu AH, Perez A, Clopton P, Krishnaswamy P, Kazanegra R, Maisel AS. B-type natriuretic peptide and clinical judgment in emergency diagnosis of heart failure: analysis from Breathing Not Properly (BNP) Multinational Study. Circulation. 2002 Jul 23;106(4):416-22. doi: 10.1161/01.cir.0000025242.79963.4c. PMID 12135939
- [Background] Moe GW, Howlett J, Januzzi JL, Zowall H; Canadian Multicenter Improved Management of Patients With Congestive Heart Failure (IMPROVE-CHF) Study Investigators. N-terminal pro-B-type natriuretic peptide testing improves the management of patients with suspected acute heart failure: primary results of the Canadian prospective randomized multicenter IMPROVE-CHF study. Circulation. 2007 Jun 19;115(24):3103-10. doi: 10.1161/CIRCULATIONAHA.106.666255. Epub 2007 Jun 4. PMID 17548729
- [Background] Steinhart B, Thorpe KE, Bayoumi AM, Moe G, Januzzi JL Jr, Mazer CD. Improving the diagnosis of acute heart failure using a validated prediction model. J Am Coll Cardiol. 2009 Oct 13;54(16):1515-21. doi: 10.1016/j.jacc.2009.05.065. PMID 19815122